CLINICAL TRIAL: NCT07404436
Title: Efficacy of Rivaroxaban for Thromboprophylaxis in Idiopathic Membranous Nephropathy: A Prospective, Single-Center, Randomized Controlled Trial
Brief Title: Rivaroxaban in Idiopathic Membranous Nephropathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Diao Zongli, Pro, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-P2-369-01
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): At present, an established rivaroxaban dosing regimen for thromboprophylaxis in IMN is lacking. In this study, we will adopt the dosing regimen used for postoperative venous thromboembolism prophylaxis (N Engl J Med, 2020, 382(20):1916-1925), administering rivaroxaban 10 mg orally once daily.
  Interventions: Drug: Rivaroxaban 10 MG
- Warfarin (Active Comparator): According to the Chinese Expert Consensus on Warfarin Anticoagulation Therapy (Chinese Journal of Internal Medicine, 2013, 52(1):76-82) and the recommendations in UpToDate (Hypercoagulability in patients with nephrotic syndrome), the protocol is as follows: Anticoagulation intensity: the target INR is 1.5-2.5. Dosing regimen: the initial warfarin dose is 1.5 mg orally once daily. INR will be measured after 3 days of treatment for inpatients or after 1 week for outpatients, and then monitored weekly thereafter. If the INR remains outside the target range on two consecutive measurements, the dose may be increased or decreased by 20% of the current dose until the INR reaches the target range.
  Interventions: Drug: Warfarin Sodium

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — At present, an established rivaroxaban dosing regimen for thromboprophylaxis in IMN is lacking. In this study, we will adopt the dosing regimen used for postoperative venous thromboembolism prophylaxis (N Engl J Med, 2020, 382(20):1916-1925), administering rivaroxaban 10 mg orally once daily.
  Arms: Rivaroxaban
Drug: Warfarin Sodium — According to the Chinese Expert Consensus on Warfarin Anticoagulation Therapy (Chinese Journal of Internal Medicine, 2013, 52(1):76-82) and the recommendations in UpToDate (Hypercoagulability in patients with nephrotic syndrome), the protocol is as follows: Anticoagulation intensity: the target INR is 1.5-2.5. Dosing regimen: the initial warfarin dose is 1.5 mg orally once daily. INR will be measured after 3 days of treatment for inpatients or after 1 week for outpatients, and then monitored weekly thereafter. If the INR remains outside the target range on two consecutive measurements, the dose may be increased or decreased by 20% of the current dose until the INR reaches the target range.
  Arms: Warfarin

SUMMARY:
Through a prospective, single-center, randomized controlled trial, we aim to determine the thromboprophylactic efficacy of rivaroxaban in patients with idiopathic membranous nephropathy (IMN). IMN patients at high risk of thrombosis and low risk of bleeding will be enrolled and randomly assigned to a rivaroxaban group or a control group (receiving warfarin). Prophylactic anticoagulation will be administered with rivaroxaban or warfarin accordingly. Over the 6 months following initiation of prophylactic anticoagulation, the incidence of the primary efficacy endpoint (a composite of pulmonary embolism, deep vein thrombosis, and lower-extremity deep vein thrombosis) and the safety endpoint (bleeding events) will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years, either sex. Kidney biopsy findings on both light microscopy and electron microscopy consistent with idiopathic membranous nephropathy (IMN).

IMN patients at high risk of thrombosis: meeting the diagnostic criteria for nephrotic syndrome and having serum albumin <25 g/L. Normal renal function (normal creatinine clearance).

Exclusion Criteria:

Prior thrombotic events, such as pulmonary embolism, renal vein thrombosis, or lower-extremity deep vein thrombosis.

Pulmonary diseases that may affect the accuracy of ventilation-perfusion (V/Q) scanning for diagnosing pulmonary embolism, such as pulmonary infection/inflammation, lung tumors, or chronic obstructive pulmonary disease.

Inability to undergo V/Q scanning, e.g., right-to-left congenital cardiac shunt, prior allergy to radiopharmaceuticals, or inability to cooperate with the examination.

Clinically significant active bleeding. Pregnant or breastfeeding women. Acute myocardial infarction and/or acute stroke, or atrial fibrillation. Active infection or active malignancy. Coagulation abnormalities; hepatic dysfunction (aminotransferases ≥3× the upper limit of normal); or thrombocytopenia (platelet count <100×10^9/L).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome | 6 months
  a composite endpoint, including the incidence of pulmonary embolism, renal vein thrombosis, and lower-extremity deep vein thrombosis.

SECONDARY OUTCOMES:
Secondary efficacy outcome | 6 months
  the incidence of pulmonary embolism, renal vein thrombosis, lower-extremity deep vein thrombosis, and other thrombotic events.

OTHER OUTCOMES:
Safety events | 6 months
  the incidence of all bleeding events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friedship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No